CLINICAL TRIAL: NCT00925353
Title: The Pharmacokinetics of 4% Lidocaine Gel When Applied Topically to the Breasts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mountain States Tumor and Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSTMRI-002
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Adverse Effects
Keywords: lidocaine; pre-medication; mammography; pain; safety
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lidocaine gel (Experimental)
  Interventions: Drug: 4% lidocaine gel

INTERVENTIONS:
Drug: 4% lidocaine gel — 1 ounce 4% lidocaine gel on skin of breasts and chest wall for 1 hour under occlusion, then removed with warm water
  Other Names: TOPICAINE

SUMMARY:
The purpose of this study is to test the hypothesis that one-time application of 4% lidocaine gel (TOPICAINE) on the skin of the breasts and chest wall as recommended for pre-medication to reduce discomfort during screening mammography does not result in adverse effects, electrocardiogram (EKG) changes, or systemically toxic plasma concentration of lidocaine or its principal metabolite, monoethylglycinexylidide (MEGX).

ELIGIBILITY:
Inclusion Criteria:

* 35 years and older
* intact skin on breasts and chest wall

Exclusion Criteria:

* sensitivity or allergy to lidocaine
* liver or kidney dysfunction
* pregnant
* breast feeding
* currently smoke or chew tobacco
* used lidocaine products within 48 hours of baseline lab, EKG, or gel application
* exhibit neurological or cardiac signs or symptoms prior to gel application
* are taking antiarrythmic medications, ciprofloxacin, erythromycin products, or oral contraceptives
* history of Wolffe-Parkinson-White Syndrome (WPW) or congestive heart failure
* heart rate below 60 or above 100 beats per minute
* systolic blood pressure below 95 or above 180 mm Hg
* PR interval greater 200 msec, QRS duration greater than 120 msec, QTc greater than 450 msec, or evidence of WPW on EKG
* have an automatic implantable cardioverter defibrillator (AICD) or cardiac pacemaker
* have had cancer, surgery, trauma, or myocardial infarction in the past 6 months

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen K Lambertz, MSN, FNP, Principal Investigator — St. Luke's Mountain States Tumor Institute
Locations (1):
- St. Luke's Mountain States Tumor Institute, Boise, Idaho, United States

REFERENCES:
- [Result] Lambertz CK, Johnson CJ, Montgomery PG, Maxwell JR, Fry SJ. Toxicity of topical lidocaine applied to the breasts to reduce discomfort during screening mammography. J Anaesthesiol Clin Pharmacol. 2012 Apr;28(2):200-4. doi: 10.4103/0970-9185.94859. PMID 22557743

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment fliers were posted at St. Luke's health System's oncology, screening mammography, internal medicine, and family health clinics, in-patient hospitals, and Boise State University.
Pre-assignment Details: 56 potential subjects responded to the fliers during the enrollment period. 31 did not meet study criteria. 13 enrolled. 3 did not meet the preliminary EKG or laboratory criteria and were withdrawn prior to gel application. 10 subjects completed the trial.
Groups:
- Lidocaine Gel: 1 ounce of lidocaine gel applied the skin of the breasts and chest wall covered by plastic wrap for one hour
Period: Overall Study
Arm/Group | Lidocaine Gel
Started | 13
Completed | 10
Not Completed | 3
Not completed — Failed preliminary EKG or lab criteria. | 3

BASELINE CHARACTERISTICS:
Arm/Group | Lidocaine Gel
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters Based on Plasma Concentration of Lidocaine and MEGX in Nanograms/Milliliter.
Description: Plasma concentration of lidocaine and MEGX in nanograms/milliliter were measured prior to one-time application of 4% lidocaine gel on the skin of the breasts and chest wall as recommended for use as as pre-medication to reduce discomfort during screening mammography, and at 30 minutes, 60 minutes, and 2, 3, 4, 6, and 8 hours. Due to the high frequency of nondetectable values, pharmacokinetic parameters could not be estimated. Measurements at all time points were grouped together to select a median.
Time Frame: Prior to gel application, and at 30 min, 60 min, and 2, 3, 4, 6, and 8 hours after
Population: Plasma lidocaine and MEGX levels were measured prior to lidociane gel application, and at 30 min, 60, min, and 2, 3, 4, 6, and 8 hours after on 10 subjects (total of 80 lidocaine levels and 80 MEGX levels). Minimum level of detection for lidocaine and MEGX was 200 ng/mL.
Measure: Median (Full Range); unit: nanograms/mililiter
Units Other Than Participants: plasma concentration
Groups:
- Lidocaine Gel Group: Plasma concentration of lidocaine and MEGX after one-time application of 1 oz. of 4% lidocaine gel (TOPICAINE) on the skin of the breasts and chest wall as recommended for use as as pre-medication to reduce discomfort during screening mammography.
Arm/Group | Lidocaine Gel Group
Number analyzed (Participants) | 10
Number analyzed (plasma concentration) | 160
nanograms/mililiter
  lidocaine | NA [NA to 310] — Measured values were below the level of detection = 200 ng/ml
  MEGX | NA [NA to NA] — Measured values were below the level of detection = 200 ng/ml
Statistical Analysis 1: Comparison: Lidocaine Gel Group; Null Hypothesis: Application of 4% lidocaine gel on the breasts and chest wall of healthy women occluded for one hour does not result in systemically toxic plasma concentrations of lidocaine or its principal metabolite, monoethylglycinexyliidie (MEGX), electrocardiogram changes, or adverse events; Test type: Superiority or Other; p < 0.05, non-compartmental pharmacokinetic; The planned analysis was to estimate pharmacokinetic parameters. There were too few detectable values to be able to perform this analysis; Actual lab results shown = 1

2. Secondary Outcome: EKG Changes
Description: The PR interval (msec), QRS duration (msec), and QTc interval (msec) were compared between the baseline and subsequent EKG using paired t-tests.
Time Frame: Prior to gel application and 3 hours after
Reporting Status: Not Posted
Measure: Mean (Standard Error); unit: msec

3. Secondary Outcome: Variation of Heart Rate (Bpm), Respiratory Rate (Respirations Per Minute, Rpm), Systolic Blood Pressure (mm Hg), and Diastolic Blood Pressure (mm Hg) Over Time.
Description: Variation of heart rate (bpm), respiratory rate (respirations per minute, rpm), systolic blood pressure (mm Hg), and diastolic blood pressure (mm Hg) over time was assessed using generalized linear mixed models with time modeled as a fixed effect and study subject modeled as a random effect.
Time Frame: Prior to gel application and at 30 min, 60 min and 2, 3, 4, 6. and 8 hours after
Reporting Status: Not Posted
Measure: Mean (Standard Error); unit: bpm, rpm, mm Hg

4. Secondary Outcome: Frequencies of Moderate, Severe, or Life-threatening Side Effects
Description: Percentages of study subjects exhibiting moderate, severe, or life-threatening signs and symptoms at each of the eight time measurements
Time Frame: Prior to gel application and at 30 min, 60 min and 2, 3, 4, 6. and 8 hours after
Reporting Status: Not Posted
Measure: Number; unit: Percentage of participants

ADVERSE EVENTS:
Arm/Group | Lidocaine Gel
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine Gel (N=10)
Skin erythema (Skin and subcutaneous tissue disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
No placebo comparison group; limited sample size; healthy subjects; lack of variation in doses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No